CLINICAL TRIAL: NCT05519839
Title: A Phase 2, Randomized, Observer-Blinded Study to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 rS Nanoparticle and Quadrivalent Hemagglutinin Nanoparticle Influenza Combination Vaccine With Matrix-M™ Adjuvant in Healthy Participants ≥ 50 to ≤ 80 Years of Age
Brief Title: A Study to Evaluate the Safety and Immunogenicity of COVID-19 and Influenza Combination Vaccine
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019nCoV-CIC-E-201
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Influenza
Keywords: Coronavirus; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human; Coronavirus Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (22):
- Group A (Part 1) (Experimental): CIC Vaccine Formulation1. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group B (Part 1) (Experimental): CIC Vaccine Formulation 2. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group C (Part 1) (Experimental): CIC Vaccine Formulation 3. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group D (Part 1) (Experimental): CIC Vaccine Formulation 3. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group E (Part 1) (Experimental): CIC Vaccine Formulation 1. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group F (Part 1) (Experimental): CIC Vaccine Formulation 2. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group G (Part 1) (Experimental): CIC Vaccine Formulation 3. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group H (Part 1) (Experimental): CIC Vaccine Formulation 4. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group I (Part 1) (Experimental): CIC Vaccine Formulation 5. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group J (Part 1) (Experimental): CIC Vaccine Formulation 6. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group K (Part 1) (Experimental): CIC Vaccine Formulation 7. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group L (Part 1) (Experimental): qNIV Vaccine Formulation 1. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: qNIV Vaccine with Matrix-M Adjuvant
- Group M (Part 1) (Experimental): qNIV Vaccine Formulation 2. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: qNIV Vaccine with Matrix-M Adjuvant
- Group N (Part 1) (Experimental): qNIV Vaccine Formulation 3 . 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: qNIV Vaccine with Matrix-M Adjuvant
- Group O (Part 1) (Experimental): SARS-CoV-2 rS Vaccine Formulation 1. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: SARS-CoV-2 rS Vaccine with Matrix-M Adjuvant
- Group P (Part 1) (Experimental): SARS-CoV-2 rS Vaccine Formulation 2. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: SARS-CoV-2 rS Vaccine with Matrix-M Adjuvant
- Group Q (Part 1) (Experimental): SARS-CoV-2 rS Vaccine Formulation 3. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: SARS-CoV-2 rS Vaccine with Matrix-M Adjuvant
- Group R (Part 1) (Experimental): SARS-CoV-2 rS Vaccine Formulation 4. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70
  Interventions: Drug: SARS-CoV-2 rS Vaccine with Matrix-M Adjuvant
- Group S (Part 1) (Experimental): Influenza Vaccine Formulation 1.
  1 intramuscular (IM) doses of vaccine, on Day 0.
  Interventions: Drug: Influenza Vaccine
- Group T (Part 2) (Experimental): CIC Vaccine Formulation 8. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70 (if applicable).
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group U (Part 2) (Experimental): CIC Vaccine Formulation 9. 2 intramuscular (IM) doses of vaccine, the first on Day 0 and the second on Day 70 (if applicable).
  Interventions: Drug: CIC Vaccine with Matrix-M Adjuvant
- Group S (Part 1)-Placebo (Placebo Comparator): 1 intramuscular (IM) doses of placebo, on Day 70.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: qNIV Vaccine with Matrix-M Adjuvant — Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV vaccine given on Day 0 and Day 70 .
  Arms: Group L (Part 1); Group M (Part 1); Group N (Part 1)
Drug: Influenza Vaccine — Intramuscular (deltoid) injections of Comparator influenza vaccine given on Day 0 and Day 70 (if applicable).
  Arms: Group S (Part 1)
Drug: CIC Vaccine with Matrix-M Adjuvant — Intramuscular (deltoid) injections of co-formulated mix of various doses and formulations of CIC Vaccine given on Day 0 and Day 70
  Arms: Group A (Part 1); Group B (Part 1); Group C (Part 1); Group D (Part 1); Group E (Part 1); Group F (Part 1); Group G (Part 1); Group H (Part 1); Group I (Part 1); Group J (Part 1); Group K (Part 1); Group T (Part 2); Group U (Part 2)
Other: Placebo Comparator — Intramuscular (deltoid) injection of placebo given on Day 70.
  Arms: Group S (Part 1)-Placebo
Drug: SARS-CoV-2 rS Vaccine with Matrix-M Adjuvant — Intramuscular (deltoid) injections of in-clinic mix of various doses of SARS-CoV-2 rS vaccine given on Day 0 and Day 70 .
  Arms: Group O (Part 1); Group P (Part 1); Group Q (Part 1); Group R (Part 1)

SUMMARY:
This is a randomized, observer-blinded, Phase 2 study evaluating the safety and immunogenicity of a severe acute respiratory syndrome coronavirus 2 (SARSCoV2) recombinant spike (rS) (SARS-CoV-2 rS) nanoparticle and quadrivalent hemagglutinin (HA) nanoparticle influenza vaccine (qNIV) combination vaccine with Matrix-M™ adjuvant; this combination vaccine.

DETAILED DESCRIPTION:
The study will enroll approximately 2300 (1520 in Part 1 and 800 in Part 2) healthy (based on history and physical examination) adult male and female participants 50 to 80 years of age, inclusive, targeting participants, who must have completed a primary vaccination series against SARS-CoV-2 with an authorized COVID-19 vaccine (and fulfill national recommendations for his/her age and morbidity category) with receipt of second/last dose of authorized vaccine (with or without boosters[s]) ≥ 3 months prior to enrollment. Randomization will be stratified by age ≥ 50 to < 65 or ≥ 65 to ≤ 80 years to distribute the proportions of each age stratum evenly across vaccine groups.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all the following criteria:

1. Medically stable adult male or females ≥ 50 to ≤ 80 years of age at screening.
2. Participants may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

   1. Absence of changes in medical therapy in the past 2 months due to treatment failure or toxicity;
   2. Absence of medical events qualifying as SAEs within 3 months; and
   3. Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the investigator.
3. The participant has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at screening.
4. Willing and able to give informed consent prior to study enrollment.
5. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AEs.
6. Participants must have completed a primary vaccination series against SARS-CoV-2 with an authorized COVID 19 vaccine (and fulfill national recommendations for his/her age and morbidity category) with receipt of second/last dose of authorized vaccine (with or without boosters[s]) ≥ 8 weeks prior to enrollment (first study vaccination).
7. Women of childbearing potential (defined as any female participant who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study

   1. Condoms (male or female) with spermicide (if acceptable in country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in-country regulatory approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle
8. Participants must be healthy and medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to vaccination.
9. Participants must agree to not participate in any other SARS-CoV-2 or influenza prevention or treatment studies for the duration of the study. Note: For participants who become hospitalized with COVID-19, participation in investigational treatment studies is permitted.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. History of laboratory-confirmed (by Polymerase Chain Reaction (PCR) or rapid antigen test) COVID-19 or asymptomatic SARS-CoV-2 infection ≤ 8 weeks prior to enrollment.

   (NOTE: Symptomatic COVID-19 or asymptomatic SARS-CoV-2 infection > 8 weeks prior to enrollment is NOT exclusionary)
2. Any ongoing, symptomatic acute illness requiring medical or surgical care or chronic illness that required changes in medication in the past 2 months indicating that chronic illness/disease is not stable (at the discretion of the investigator). This includes any current workup of undiagnosed illness that could lead to a new condition.
3. Serious chronic diseases inclusive of:

   1. Uncontrolled hypertension (NOTE: well controlled hypertension ≤ grade 2 in NOT exclusionary);
   2. Congestive heart failure with a history of an acute exacerbation of any severity in the prior 2 years (NOTE:

      mild well-controlled congestive heart failure is NOT exclusionary);
   3. Chronic obstructive pulmonary disease (COPD) with a history of an acute exacerbation of any severity in the prior 2 years (NOTE: mild well-controlled COPD is NOT exclusionary);
   4. In the past 3 months, evidence of unstable coronary artery disease as manifested by cardiac interventions (eg, cardiac stent placement, coronary artery bypass grafting [CABG]) surgery, new cardiac medications for control of symptoms, or unstable angina (NOTE: stable coronary heart disease is NOT exclusionary);
   5. Asthma with a history of exacerbation in the prior 2 years or worsening of asthma symptoms or requiring changes in asthma control medications in the past 2 months (NOTE: well-controlled asthma is NOT exclusionary).
   6. Type 1 or type 2 diabetes (adult onset) requiring insulin (NOTE: non-insulin dependent type 2 diabetes is NOT exclusionary);
   7. Chronic kidney disease/renal insufficiency;
   8. Chronic gastrointestinal and hepatic diseases; or
   9. Chronic neurological diseases (such as multiple sclerosis, dementia, Parkinson's disease, degenerative neurological conditions, neuropathy, or epilepsy), history of stroke within 12 months with residual symptoms, or previous neurological disorder within 12 months with residual symptoms (NOTE: history of migraine or chronic headaches or nerve root compression that have been stable on treatment for the last 4 weeks are NOT exclusionary).
4. Participation in research involving an investigational product (drug/biologic/device) within 90 days before planned date of vaccination.
5. Use of COVID-19 prophylactic or treatment monoclonal antibodies or antibody cocktails within 90 days prior to planned date of vaccination.
6. History of a serious reaction to prior influenza vaccination or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80; or any known allergies to products contained in the investigational product.
7. Any history of anaphylaxis to any prior vaccine.
8. History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine.
9. Receipt of any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within 8 weeks preceding the study vaccination. Note: Routine vaccinations will not be allowed until after study Day 21 and COVID and influenza vaccination will not be allowed until after Day 84.
10. Any known or suspected autoimmune or immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination (NOTE: mild psoriasis is not exclusionary).
11. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune- modifying drugs within 6 months prior to the administration of the study vaccines. An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted.
12. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
13. Active cancer (malignancy) therapy within 3 years prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
14. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study (EoS).
15. Known disturbance of coagulation.
16. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination, which in the opinion of the investigator, might interfere with protocol compliance.
17. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature > 38.0°C, on the planned day of vaccine administration).
18. History of myocarditis or pericarditis.
19. Any condition that in the opinion of the investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
20. Study team member or immediate family member of any study team member (inclusive of Sponsor, Contract Research Organization, and study site personnel involved in the conduct or planning of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1579 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2 : Number of participants with solicited local and systemic Adverse Events (AEs) | Day 0 to Day 7
  Numbers of participants with solicited local and systemic AEs over the 7 days post-vaccination.
Part 1 and Part 2 : Percentage of participants with all AEs | Day 0 to Day 21
  Proportions of participants reporting all AEs, solicited and unsolicited, over 21 days post-vaccination.
Part 1 and Part 2 : Percentage of participants with Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs) | Day 0 to Day 182
  Proportions of participants with MAAEs, AESIs (including PIMMCs and myocarditis and/or pericarditis), SAEs, will be collected for 6 months (approximately 182 days) post-vaccination

SECONDARY OUTCOMES:
Part 1 and Part 2 : Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and Antigenically Drifted Influenza Strains Expressed as Geometric Mean Titer (GMT) | Day 0 to Day 84
  HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s), and antigenically drifted influenza strains. Derived/calculated endpoints based on GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 0, 7, 21, 84, and other follow-up time points
Part 1 and Part 2 : Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and Antigenically Drifted Influenza Strains Expressed as Geometric Mean Fold Rise (GMFR) | Day 0 to Day 84
  HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s), and antigenically drifted influenza strains. Derived/calculated endpoints based on Geometric mean fold rise (GMFRPost/Pre) - defined as the within group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 7, 21, 84, and other follow-up time points.
Part 1 and Part 2 : Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and Antigenically Drifted Influenza Strains Expressed as Seroconversion Rate (SCR) | Day 0 to Day 84
  HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s), and antigenically drifted influenza strains. Derived/calculated endpoints based on Seroconversion rate (SCR) - defined as proportion of participants in a given Vaccine Group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 7, 21, 84, and other follow-up time points
Part 1 and Part 2 : Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and Antigenically Drifted Influenza Strains Expressed as Seroprotection Rate (SPR) | Day 0 to Day 84
  HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s), and antigenically drifted influenza strains. Derived/calculated endpoints based on Seroprotection rate (SPR) - defined as the proportion of participants with a reciprocal HAI titer ≥ 40 on Days 7, 21, 84, and other follow-up time points.
Part 1 and Part 2 : Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and Antigenically Drifted Influenza Strains Expressed as Geometric Mean Titer Ratio (GMTR) | Day 0 to Day 84
  HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s), and antigenically drifted influenza strains. Derived/calculated endpoints based on GMTR between select treatment arms at Days 7, 21, 84, and other follow-up time points post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers).
Part 1 and Part 2: Neutralizing Antibody Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and/or Antigenically Drifted Influenza Strains Expressed as GMTs | Day 0 to Day 84
  Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B strain(s) and/or antigenically drifted influenza strains, as measured by a MN assay expressed as GMTs.
Part 1 and Part 2 : Neutralizing Antibody Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and/or Antigenically Drifted Influenza Strains Expressed as GMFR | Day 0 to Day 84
  Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B strain(s) and/or antigenically drifted influenza strains, as measured by a MN assay expressed as GMFR
Part 1 and Part 2: Neutralizing Antibody Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and/or Antigenically Drifted Influenza Strains Expressed as SCR | Day 0 to Day 84
  Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B strain(s) and/or antigenically drifted influenza strains, as measured by a MN assay expressed as SCR.
Part 1 and Part 2: Neutralizing Antibody Titers Specific for Vaccine Homologous A and B Influenza Strain(s) and/or Antigenically Drifted Influenza Strains Expressed as GMTR | Day 0 to Day 84
  Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B strain(s) and/or antigenically drifted influenza strains, as measured by a MN assay expressed as GMTR.
Part 1 and Part 2: Serum Immunoglobulin G (IgG) to the SARS-CoV-2 spike protein expressed as GMEU | Day 0 to Day 84
  IgG geometric mean enzyme-linked immunosorbent assay (ELISA) unit (GMEU) concentrations (EU/mL) to the SARS-CoV-2 S protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points, expressed as GMEU.
Part 1 and Part 2: Serum IgG to the SARS-CoV-2 spike protein expressed as GMFR | Day 0 to Day 84
  IgG geometric mean enzyme-linked immunosorbent assay (ELISA) unit (GMEU) concentrations (EU/mL) to the SARS-CoV-2 S protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points, expressed as GMFR.
Part 1 and Part 2: Serum IgG to the SARS-CoV-2 spike protein expressed as SCR | Day 0 to Day 84
  IgG geometric mean enzyme-linked immunosorbent assay (ELISA) unit (GMEU) concentrations (EU/mL) to the SARS-CoV-2 S protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points expressed as SCR.
Part 1 and Part 2: Serum IgG to the SARS-CoV-2 spike protein expressed as Geometric Mean ELISA Unit Ratio (GMEUR) | Day 0 to Day 84
  IgG geometric mean enzyme-linked immunosorbent assay (ELISA) unit (GMEU) concentrations (EU/mL) to the SARS-CoV-2 S protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points, expressed as GMEUR.
Part 1 and Part 2: Microneutralization assay (MN) 50 GMTs to the SARS-CoV-2 expressed as GMTs | Day 0 to Day 84
  MN50 GMTs to the SARS-CoV-2 from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points, expressed as GMTs.
Part 1 and Part 2: MN50 GMTs to the SARS-CoV-2 expressed as GMFR | Day 0 to Day 84
  MN50 GMTs to the SARS-CoV-2 from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points expressed as GMFR.
Part 1 and Part 2: MN50 GMTs to the SARS-CoV-2 expressed as SCR | Day 0 to Day 84
  MN50 GMTs to the SARS-CoV-2 from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points expressed as SCR.
Part 1 and Part 2: MN50 GMTs to the SARS-CoV-2 expressed as GMTR | Day 0 to Day 84
  MN50 GMTs to the SARS-CoV-2 from the matched vaccine construct (and mismatched variant if available), at Days 0, 7, 21, 84, and other follow-up time points expressed as GMTR

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (35):
- Australia (25):
  - Paratus Clinical Research - Canberra, Bruce, Australian Capital Territory
  - Paratus Clinical Research - Western Sydney, Blacktown, New South Wales
  - Emeritus Research - Sydney, Botany, New South Wales
  - Genesis Central Coast, Broadmeadow, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Holdsworth House Medical Brisbane, Darlinghurst, New South Wales
  - Oztrials Clinical Research, Drummoyne, New South Wales
  - Paratus Clinical Research - Central Coast, Kanwal, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Sutherland Clinical Trials, Miranda, New South Wales
  - Illawarra Health and Medical Research Institute, Wollongong, New South Wales
  - Northside Health, Coffs Harbour, New South Whales
  - Novatrials, Kotara, New South Whales
  - Menzies Darwin, Tiwi, Norther Territory
  - Paratus Clinical Research - Brisbane Clinic, Albion, Queensland
  - Mater Adult Hospital, Brisbane, Queensland
  - Nucleus Network Pty Ltd, Herston, Queensland
  - Core Research Group, Milton, Queensland
  - Austrials Pty Ltd - Taringa, Taringa, Queensland
  - AusTrials (Wellers Hill), Tarragindi, Queensland
  - CMAX, Adelaide, South Australia
  - Emeritus Research, Camberwell, Victoria
  - Nucleus Network Limited, Melbourne, Victoria
- New Zealand (10):
  - P3 Reseach - Hawkes Bay, Havelock North, Hawkes Bay
  - P3 Research - Palmerston North, Palmerston North, Manawatu-Wanganui
  - P3 Research - Lower Hutt, Palmerston, Wellington Region
  - P3 Research Kapiti, Paraparaumu, Wellington Region
  - Middlemore Clinical Trials, Auckland
  - Optimal Clinical Trials Ltd, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch
  - P3 Research - Dunedin, Dunedin
  - P3 Research - Tauranga, Tauranga
  - P3 Research - Wellington, Wellington